CLINICAL TRIAL: NCT02614287
Title: A Phase 3, Long-Term, Open-Label Safety Study of LY2951742 in Patients With Migraine
Brief Title: A Safety Study of Galcanezumab in Participants With Migraine, With or Without Aura
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15770; I5Q-MC-CGAJ (Other: Eli Lilly and Company); 2015-001884-38 (EudraCT Number)
Record Dates: First submitted 2015-11-23; First posted 2015-11-25 (Estimated); Results first posted 2019-01-07 (Actual); Last update posted 2020-06-17 (Actual); Status verified 2020-06

CONDITIONS: Migraine
Keywords: prevention; prophylaxis; headache
MeSH Terms: conditions — Migraine Disorders; Headache | interventions — galcanezumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Galcanezumab 120 mg (Experimental): Galcanezumab 240mg given as loading dose at first dosing visit followed by 120 mg given by subcutaneous (SC) injection once a month for up to 11 months by auto injector or pre-filled syringe.
  Interventions: Drug: Galcanezumab
- Galcanezumab 240 mg (Experimental): Galcanezumab 240 mg given by SC injection once a month for up to 12 months by auto injector or pre-filled syringe.
  Interventions: Drug: Galcanezumab

INTERVENTIONS:
Drug: Galcanezumab — Administered SC
  Other Names: LY2951742

SUMMARY:
The main purpose of this study is to evaluate the longer term safety of the study drug known as galcanezumab in participants with episodic or chronic migraine.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of episodic or chronic migraine as defined by International Headache Society (IHS) International Classification of Headache Disorders (ICHD)-3 beta guidelines (1.1, 1.2 or 1.3) (ICHD-3 2013), with a history of migraine headaches of at least 1 year prior to screening, and migraine onset prior to age 50.
* Prior to baseline, a history of 4 or more migraine headache days per month on average for the past 3 months.

Exclusion Criteria:

* Are currently enrolled in or have participated within the last 30 days or within 5 half-lives (whichever is longer) in a clinical trial involving an investigational product.
* Current use or prior exposure to galcanezumab or another CGRP antibody.
* Known hypersensitivity to multiple drugs, monoclonal antibodies or other therapeutic proteins, or to galcanezumab.
* History of persistent daily headache, cluster headache or migraine subtypes including hemiplegic (sporadic or familial) migraine, ophthalmoplegic migraine, and migraine with brainstem aura (basilar-type migraine) defined by IHS ICHD-3 beta.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Actual)
Dates: Start 2015-11-30 (Actual); Primary Completion 2017-05-12 (Actual); Study Completion 2018-08-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (27):
- United States (13):
  - California Medical Clinic for Headache, Santa Monica, California
  - Encompass Clinical Research, Spring Valley, California
  - New England Institute for Clinical Research, Stamford, Connecticut
  - Sunrise Clinical Research, Hollywood, Florida
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - Mercy Health Research, St Louis, Missouri
  - Albuquerque Neurosciences, Albuquerque, New Mexico
  - PharmQuest, Greensboro, North Carolina
  - Wilmington Health Associates, Wilmington, North Carolina
  - Suburban Research Associates, Media, Pennsylvania
  - Clinpoint Trial, LLC, Waxahachie, Texas
  - Ericksen Research and Development, Clinton, Utah
  - Blue Ridge Research Center, Roanoke, Virginia
- Belgium (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bruges
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Brussels
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Liège
- Canada (3):
  - For additional information regarding investigative sites for this trial, contact 1-888-545-5972 Mon - Fri, 9 AM to 4 PM or 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time or speak with your personal physician., Calgary
  - For additional information regarding investigative sites for this trial, contact 1-888-545-5972 Mon - Fri, 9 AM to 4 PM or 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time or speak with your personal physician., Sherbrooke
  - For additional information regarding investigative sites for this trial, contact 1-888-545-5972 Mon - Fri, 9 AM to 4 PM or 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time or speak with your personal physician., Toronto
- France (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Marseille
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nice
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Paris
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saint-Etienne
- Hungary (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Budapest
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Esztergom
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Győr
- Ponce School of Medicine CAIMED Center, Ponce, Puerto Rico

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- [Derived] Stauffer VL, Turner I, Kemmer P, Kielbasa W, Day K, Port M, Quinlan T, Camporeale A. Effect of age on pharmacokinetics, efficacy, and safety of galcanezumab treatment in adult patients with migraine: results from six phase 2 and phase 3 randomized clinical trials. J Headache Pain. 2020 Jun 23;21(1):79. doi: 10.1186/s10194-020-01148-9. PMID 32576229
- [Derived] Bangs ME, Kudrow D, Wang S, Oakes TM, Terwindt GM, Magis D, Yunes-Medina L, Stauffer VL. Safety and tolerability of monthly galcanezumab injections in patients with migraine: integrated results from migraine clinical studies. BMC Neurol. 2020 Jan 17;20(1):25. doi: 10.1186/s12883-020-1609-7. PMID 31952501
- [Derived] Kielbasa W, Quinlan T. Population Pharmacokinetics of Galcanezumab, an Anti-CGRP Antibody, Following Subcutaneous Dosing to Healthy Individuals and Patients With Migraine. J Clin Pharmacol. 2020 Feb;60(2):229-239. doi: 10.1002/jcph.1511. Epub 2019 Sep 4. PMID 31482569
- [Derived] Camporeale A, Kudrow D, Sides R, Wang S, Van Dycke A, Selzler KJ, Stauffer VL. A phase 3, long-term, open-label safety study of Galcanezumab in patients with migraine. BMC Neurol. 2018 Nov 9;18(1):188. doi: 10.1186/s12883-018-1193-2. PMID 30413151
- See also: Click here for more information about this study: A Safety Study of Galcanezumab in Participants With Migraine, With or Without Aura — http://www.lillytrialguide.com/EN-US/studies/headache/cgaj

RESULTS

PARTICIPANT FLOW:
Groups:
- Galcanezumab 120 mg: Participants received a loading dose of 240 milligram (mg) galcanezumab at first dosing visit followed by120 mg galcanezumab once a month by subcutaneous injection during open label treatment phase. Participants did not receive any intervention during post treatment follow-up phase.
- Galcanezumab 240 mg: Participants received 240 mg of galcanezumab once a month by subcutaneous injection during open label treatment phase. Participants did not receive any intervention during post treatment follow-up phase.
Period: Open Label (OL) Treatment Phase
Arm/Group | Galcanezumab 120 mg | Galcanezumab 240 mg
Started | 135 | 135
Received at Least One Dose of Study Drug | 135 | 135
Completed | 97 | 113
Not Completed | 38 | 22
Not completed — Adverse Event | 7 | 6
Not completed — Lack of Efficacy | 13 | 5
Not completed — Lost to Follow-up | 7 | 4
Not completed — Physician Decision | 1 | 0
Not completed — Withdrawal by Subject | 10 | 7
Period: Post Treatment Follow-up Phase
Arm/Group | Galcanezumab 120 mg | Galcanezumab 240 mg
Started | 112 (Follow-up period was optional, few participants who completed OL period didn't enter follow-up.) | 124 (Follow-up period was optional, few participants who completed OL period didn't enter follow-up.)
Completed | 103 | 119
Not Completed | 9 | 5
Not completed — Adverse Event | 1 | 0
Not completed — Lost to Follow-up | 2 | 2
Not completed — Withdrawal by Subject | 6 | 3

BASELINE CHARACTERISTICS:
Population: All randomized participants
Groups:
- Galcanezumab 120 mg: Participants received a loading dose of 240 mg galcanezumab at first dosing visit followed by 120 mg galcanezumab once a month by subcutaneous injection during open label treatment phase & participants did not receive any intervention during post treatment follow-up phase.
- Galcanezumab 240 mg: Participants received 240 mg galcanezumab once a month by subcutaneous injection during open label treatment phase & participants did not receive any intervention during post treatment follow-up phase.
- Total: Total of all reporting groups
Arm/Group | Galcanezumab 120 mg | Galcanezumab 240 mg | Total
Number analyzed (Participants) | 135 | 135 | 270
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.21 (11.68) | 43.69 (10.99) | 41.95 (11.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 110 | 113 | 223
  Male | 25 | 22 | 47
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: All randomized participants with ethnicity data.
  Participants
    number analyzed (Participants) | 127 | 128 | 255
    Hispanic or Latino | 12 | 20 | 32
    Not Hispanic or Latino | 115 | 108 | 223
    Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 6 | 8 | 14
  White | 103 | 108 | 211
  More than one race | 23 | 19 | 42
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Discontinued Due to Adverse Event
Description: Adverse Event: Any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product that does not necessarily have a causal relationship with this treatment. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product.
  A summary of other non-serious AEs, and all SAE's, regardless of causality, is reported in the Adverse Events section.
Time Frame: Baseline through Month 12
Population: All randomized participants who received at least one dose of study drug. There were 6 participants in the 120 mg group who discontinued after receiving loading dose of 240mg, these participants were moved to 240mg group for AE analysis.
Measure: Number; unit: Percentage of Participants
Groups:
- Galcanezumab 120 mg: Participants received a loading dose of 240 mg galcanezumab at first dosing visit followed by 120 mg galcanezumab once a month by subcutaneous injection 11 months.
- Galcanezumab 240 mg: Participants received 240 mg of galcanezumab once a month by subcutaneous injection for 12 months.
Arm/Group | Galcanezumab 120 mg | Galcanezumab 240 mg
Number analyzed (Participants) | 129 | 141
Percentage of Participants | 4.65 | 4.96
Statistical Analysis 1: Comparison: Galcanezumab 120 mg vs Galcanezumab 240 mg; Test type: Superiority; p = 1, Fisher Exact

2. Secondary Outcome: Pharmacokinetics (PK): Area Under the Concentration Time Curve (AUC) of Galcanezumab
Description: Pharmacokinetics (PK): Area Under the Concentration Time Curve (AUC) of Galcanezumab
Time Frame: Baseline through Month 12
Population: Zero participants analyzed. AUC data was not collected as AUC was not pre-specified in protocol.
Groups:
- Galcanezumab 120 mg: Participants received a loading dose of 240 mg galcanezumab at first dosing visit followed by 120 mg galcanezumab once a month by subcutaneous injection for 11 months.
Arm/Group | Galcanezumab 120 mg | Galcanezumab 240 mg
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Serum Concentrations of Galcanezumab
Description: Serum Concentrations of Galcanezumab.
Time Frame: Month 12
Population: All randomized participants with measurable serum concentrations at month 12.
Measure: Mean (Standard Deviation); unit: Nanogram per milliliter (ng/mL)
Groups:
- Galcanezumab 120 mg: Participants received a loading dose of 240 mg galcanezumab at first dosing visit followed by 120 mg galcanezumab once a month by subcutaneous injection for 12 months.
Arm/Group | Galcanezumab 120 mg | Galcanezumab 240 mg
Number analyzed (Participants) | 61 | 78
Nanogram per milliliter (ng/mL) | 16500 (8370) | 31600 (15900)

4. Secondary Outcome: Plasma Concentration of Calcitonin Gene-Related Peptide (CGRP)
Description: Plasma Concentration of Calcitonin Gene-Related Peptide (CGRP)
Time Frame: Month 12
Population: All randomized participants with measurable plasma concentration.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Galcanezumab 120 mg | Galcanezumab 240 mg
Number analyzed (Participants) | 87 | 103
ng/mL | 2.74 (1.07) | 3.85 (1.85)

5. Secondary Outcome: Percentage of Participants Developing Anti-Drug Antibodies to Galcanezumab
Description: A Treatment Emergent Anti-drug Antibody (TE ADA) evaluable participant is considered to be TE ADA+ if the participant has at least one post-baseline titer that is a 4-fold or greater increase in titer from baseline measurement. If baseline result is ADA Not Present, then the participant is TE ADA+ if there is at least one post-baseline result of ADA Present with titer >= 1: 20 (treatment-induced).
  There were 6 participants in the 120 mg arm who discontinued after receiving loading dose of 240mg, these participants were moved to 240mg arm for safety analysis.
Time Frame: Month 1 through Month 12
Population: All randomized participants who received at least one dose of study drug and had baseline and at least one post baseline evaluable data for TE ADA.
Measure: Number; unit: Percentage of Participants
Arm/Group | Galcanezumab 120 mg | Galcanezumab 240 mg
Number analyzed (Participants) | 129 | 137
Percentage of Participants | 12.40 | 7.30
Statistical Analysis 1: Comparison: Galcanezumab 120 mg vs Galcanezumab 240 mg; TE ADA Positive (TE ADA+); Test type: Superiority; p = .215, Fisher Exact

6. Secondary Outcome: Overall Mean Change From Baseline in the Number of Migraine Headache Days (MHD)
Description: MHD: A calendar day on which a migraine headache or probable migraine headache occurred. Overall mean is derived from the average of months 1 to 12 from MMRM model. Least squares mean (LSMean) was calculated using mixed model repeated measures (MMRM) model with treatment, pooled investigative site, month, and treatment by month, baseline, and baseline by month as fixed effects.
Time Frame: Baseline, Month 1 through Month 12
Population: All randomized participants who received at least one dose of study drug and had baseline & at least one post baseline value.
Measure: Least Squares Mean (Standard Error); unit: Migraine Headache Days per Month
Arm/Group | Galcanezumab 120 mg | Galcanezumab 240 mg
Number analyzed (Participants) | 132 | 135
Migraine Headache Days per Month | -5.61 (0.34) | -6.47 (0.33)
Statistical Analysis 1: Comparison: Galcanezumab 120 mg vs Galcanezumab 240 mg; Test type: Superiority; p = 0.60, Mixed Models Analysis; LSMean Difference = -0.86, 95% CI 2-sided [-1.76 to 0.04], Standard Error of Mean 0.46

7. Secondary Outcome: Overall Mean Change From Baseline in the Number of Headache Days
Description: Headache Day: A calendar day on which any type of headache occurred (including migraine, probable migraine, and non-migraine headache).
  Overall mean is derived from the average of months 1 to 12 from MMRM model. LSMean was calculated using MMRM model with treatment, pooled investigative site, month, and treatment by month, baseline, and baseline by month as fixed effects.
Time Frame: Baseline, Month 1 through Month 12
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: Headache Days per Month
Arm/Group | Galcanezumab 120 mg | Galcanezumab 240 mg
Number analyzed (Participants) | 132 | 135
Headache Days per Month | -2.17 (0.30) | -2.09 (0.30)
Statistical Analysis 1: Comparison: Galcanezumab 120 mg vs Galcanezumab 240 mg; Test type: Superiority; p = .835, Mixed Models Analysis; LSMean Difference = 0.09, 95% CI 2-sided [-0.72 to 0.89], Standard Error of Mean 0.41

8. Secondary Outcome: Percentage of Participants With Overall Reduction From Baseline ≥50% in Monthly Migraine Headache Days
Description: Migraine Headache Day: A calendar day on which a migraine headache or probable migraine headache occurred.
  Overall percentage of participants with a given response rate were estimated from the generalized linear mixed models (GLIMMIX) model.
Time Frame: Baseline, Month 1 through Month 12
Population: as for outcome 6
Measure: Number; unit: percentage of Participants
Arm/Group | Galcanezumab 120 mg | Galcanezumab 240 mg
Number analyzed (Participants) | 95 | 112
percentage of Participants | 65.6 | 73.7
Statistical Analysis 1: Comparison: Galcanezumab 120 mg vs Galcanezumab 240 mg; Test type: Superiority; p = .063, CPLRM; CPLRM: Categorical pseudo likelihood-based repeated measures model; Odds Ratio (OR) = 1.467, 95% CI 2-sided [0.979 to 2.197]

9. Secondary Outcome: Overall Mean Change From Baseline in the Frequency of Medication Use for the Acute Treatment of Migraines or Headaches
Description: Overall mean is derived from the average of months 1 to 12 from MMRM model. LSMean was calculated using MMRM model with treatment, pooled investigative site, month, and treatment by month, baseline, and baseline by month as fixed effects.
Time Frame: Baseline, Month 1 through Month 12
Population: All randomized participants who received at least one dose of study drug and had baseline and at least one post baseline value.
Measure: Least Squares Mean (Standard Error); unit: Medication Used Days per Month
Arm/Group | Galcanezumab 120 mg | Galcanezumab 240 mg
Number analyzed (Participants) | 132 | 135
Medication Used Days per Month | -5.09 (0.38) | -5.05 (0.37)
Statistical Analysis 1: Comparison: Galcanezumab 120 mg vs Galcanezumab 240 mg; Test type: Superiority; p = .937, Mixed Models Analysis; LSMean Difference = 0.04, 95% CI 2-sided [-0.96 to 1.04], Standard Error of Mean 0.51

10. Secondary Outcome: Overall Mean Patient Global Impression-Improvement (PGI-I) Score
Description: The Patient Global Impression of Improvement (PGI -I) scale is a participant-rated instrument that measures the participants own global impression of their symptom improvement. The participant was instructed as follows: "Mark the box that best describes your migraine headache condition since you started taking this medicine." Response options were on a 7-point scale in which a score of 1 indicates that the participant's condition is "very much better," a score of 4 indicates that the participant has experienced "no change," and a score of 7 indicates that the participant is "very much worse." Overall mean is derived from the average of months 1 to 12 from MMRM model. LSMean was calculated using MMRM model with treatment, pooled investigative site, month, and treatment by month, baseline PGI-S, and baseline PGI-S by month as fixed effects.
Time Frame: Month 1 through Month 12
Population: All randomized participants who received at least one dose of study drug and had at least one post baseline value.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Galcanezumab 120 mg | Galcanezumab 240 mg
Number analyzed (Participants) | 130 | 135
units on a scale | 2.18 (0.08) | 1.99 (0.08)
Statistical Analysis 1: Comparison: Galcanezumab 120 mg vs Galcanezumab 240 mg; Test type: Superiority; p = 0.073, Mixed Models Analysis; LSMean Difference = -0.19, 95% CI 2-sided [-0.40 to 0.02], Standard Error of Mean 0.10

11. Secondary Outcome: Overall Mean Change From Baseline on the Migraine Disability Assessment Test (MIDAS) Total Score
Description: The MIDAS is a participant-rated scale which was designed to quantify headache-related disability over a 3-month period. This instrument consists of five items that reflect the number of days reported as missing or with reduced productivity at work or home, and the number of days of missed social events. Each item has a numeric response range from 0 to 90 days, if days are missed from work or home they are not counted as days with reduced productivity at work or home. The numeric responses are summed to produce a total score ranging from 0 to 270, in which a higher value is indicative of more disability. Overall mean is derived from the average of months 1 to 12 from MMRM model. LSMean was calculated using MMRM model with treatment, pooled investigative site, month, and treatment by month, baseline, and baseline by month.
Time Frame: Baseline, Month 1 through Month 12
Population: as for outcome 9
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- Galcanezumab 120 mg: Participants received a loading dose of 240 mg of galcanezumab at first dosing visit followed by 120 mg galcanezumab once a month by subcutaneous injection for 11 months.
Arm/Group | Galcanezumab 120 mg | Galcanezumab 240 mg
Number analyzed (Participants) | 124 | 130
units on a scale | -33.58 (2.11) | -32.67 (2.04)
Statistical Analysis 1: Comparison: Galcanezumab 120 mg vs Galcanezumab 240 mg; Test type: Superiority; p = .747, Mixed Models Analysis; LSMean Difference = 0.91, 95% CI 2-sided [-4.65 to 6.47], Standard Error of Mean 2.82

12. Secondary Outcome: Overall Mean Change From Baseline on the Migraine-Specific Quality of Life Questionnaire (MSQ) Version 2.1
Description: MSQv2.1 is a health status instrument,with a 4-week recall period, developed to address physical & emotional limitations of specific concern to individuals with migraine. Addressing the impact of migraine on work or daily activities, relationships with family & friends, leisure time, productivity, concentration, energy, tiredness & feelings.It consists of 14 items addressing 3 domains:(1)Role Function-Restrictive (items 1-7);(2)Role Function- Preventive (items 8-11);&(3)Emotional Function (items 12-14).Response options range from "none of the time" (value 1) to "all of the time" (value 6), & are reverse-recoded (value 6 to 1) before the domain scores are calculated. Total raw scores for each domain is the sum of the final item value for all of the items in that domain.After total raw score is computed for each domain & total score, they are transformed to a 0-100 scale with higher scores indicating a better health status & a positive change in scores reflecting functional improvement.
Time Frame: Baseline, Month 1 through Month 12
Population: All randomized participants who received at least one dose of study drug and had baseline and at least one post baseline value.
  Overall mean is derived from the average of months 1 to 12.LSMean was calculated using MMRM model with treatment, pooled investigative site, month, and treatment by month, baseline, and baseline by month as fixed effects.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Galcanezumab 120 mg | Galcanezumab 240 mg
Number analyzed (Participants) | 130 | 135
units on a scale
  Total Score | 28.27 (1.16) | 30.25 (1.13)
  Role Function-Restrictive Domain | 31.55 (1.20) | 33.40 (1.16)
  Role Function-Preventive Domain | 22.08 (1.11) | 23.33 (1.08)
  Emotional Function Domain | 28.92 (1.35) | 32.01 (1.31)
Statistical Analysis 1: Comparison: Galcanezumab 120 mg vs Galcanezumab 240 mg; Total Score; Test type: Superiority; p = 0.203, Mixed Models Analysis; LSMean Difference = 1.98, 95% CI 2-sided [-1.07 to 5.03], Standard Error of Mean 1.55
Statistical Analysis 2: Comparison: Galcanezumab 120 mg vs Galcanezumab 240 mg; Role Function-Restrictive Domain Score; Test type: Superiority; p = .247, Mixed Models Analysis; LSMean Difference = 1.85, 95% CI 2-sided [-1.29 to 4.98], Standard Error of Mean 1.59
Statistical Analysis 3: Comparison: Galcanezumab 120 mg vs Galcanezumab 240 mg; Role Function-Preventive Domain Score; Test type: Superiority; p = 0.399, Mixed Models Analysis; LSMean Difference = 1.26, 95% CI 2-sided [-1.67 to 4.19], Standard Error of Mean 1.49
Statistical Analysis 4: Comparison: Galcanezumab 120 mg vs Galcanezumab 240 mg; Emotional Function Domain Score; Test type: Superiority; p = 0.88, Mixed Models Analysis; LSMean Difference = 3.09, 95% CI 2-sided [-0.46 to 6.64], Standard Error of Mean 1.80

13. Secondary Outcome: Percentage of Participants With Positive Responses on Patient Satisfaction With Medication Questionnaire-Modified (PSMQ-M)
Description: The PSMQ-M is a self-rated scale which measures participants level of satisfaction with study medication.The scale has been modified for use in this study, assessing 3 items related to the clinical trial treatment over the past 4 weeks: satisfaction, preference, and side effects. Satisfaction responses range from "very unsatisfied" to "very satisfied" with the current treatment. Preference compares the current study medication to previous medications, with responses from "much rather prefer my previous medication" to "much rather prefer the medication administered to me during the study".
Time Frame: Baseline through Month 12
Population: All randomized participants who received at least one dose of study drug and had month 12 PSMQ-M measurement.
Measure: Number; unit: percentage of Participants
Arm/Group | Galcanezumab 120 mg | Galcanezumab 240 mg
Number analyzed (Participants) | 90 | 112
percentage of Participants
  Satisfaction: Very satisfied | 57.78 | 58.04
  Satisfaction: Somewhat satisfied | 18.89 | 15.18
  Preference: Much prefer study medication | 66.67 | 63.39
  Preference: Prefer study medication | 22.22 | 17.86
  Side effects: Much less side effects | 66.67 | 50.89
  Side effects: Less side effects | 14.44 | 30.36

14. Secondary Outcome: Number of Participant Visits With Positive Reponses by Device Type Subcutaneous Administration Assessment Questionnaire Q1, Q3-Q12
Description: The SQAAQ is a self-administered questionnaire that provides an assessment of ease of use and confidence with using a device to administer a subcutaneous injection of study drug. Participants will respond to questionnaire items using a 7-point Likert scale (from "Strongly Disagree" to "Strongly Agree") shortly after the injection. If a caregiver administers the injection, the participants should be prepared to provide the caregiver's ratings of the questions.strongly agree & agree are considered as positive responses.
Time Frame: Baseline through Month 12
Population: All randomized participants who switched from pre-filled syringe and received at least one dose of study drug by autoinjector.
Measure: Number; unit: participants
Units Other Than Participants: Number of participant visits
Arm/Group | Galcanezumab 120 mg | Galcanezumab 240 mg
Number analyzed (Participants) | 84 | 95
Number analyzed (Number of participant visits) | 899 | 1032
participants
  Pre-filled Syringe : Easy to learn how to use: number analyzed (Number of participant visits) | 646 | 751
  Pre-filled Syringe : Easy to learn how to use | 611 | 688
  Pre-filled Syringe : Easy to hold in hand: number analyzed (Number of participant visits) | 646 | 751
  Pre-filled Syringe : Easy to hold in hand | 589 | 660
  Pre-filled Syringe : Easy to inject my dose: number analyzed (Number of participant visits) | 645 | 751
  Pre-filled Syringe : Easy to inject my dose | 580 | 659
  Pre-filled Syringe : Easy to know dose is complete: number analyzed (Number of participant visits) | 646 | 751
  Pre-filled Syringe : Easy to know dose is complete | 615 | 703
  Pre-filled Syringe: Easy to store device in fridge: number analyzed (Number of participant visits) | 625 | 726
  Pre-filled Syringe: Easy to store device in fridge | 536 | 630
  Pre-filled Syringe : Easy to remove needle shield: number analyzed (Number of participant visits) | 646 | 751
  Pre-filled Syringe : Easy to remove needle shield | 610 | 699
  Pre-filled Syringe : Easy to pickup: number analyzed (Number of participant visits) | 646 | 751
  Pre-filled Syringe : Easy to pickup | 610 | 693
  Pre-filled Syringe : overall, easy to use: number analyzed (Number of participant visits) | 646 | 751
  Pre-filled Syringe : overall, easy to use | 600 | 663
  Pre-filled Syringe:Dvc is stable against skin: number analyzed (Number of participant visits) | 646 | 744
  Pre-filled Syringe:Dvc is stable against skin | 590 | 652
  Pre-filled Syringe:Confident in ability to use: number analyzed (Number of participant visits) | 646 | 751
  Pre-filled Syringe:Confident in ability to use | 580 | 654
  Pre-filled Syringe : Confident my dose is complete: number analyzed (Number of participant visits) | 646 | 751
  Pre-filled Syringe : Confident my dose is complete | 618 | 708
  Autoinjector : Easy to learn how to use: number analyzed (Number of participant visits) | 253 | 281
  Autoinjector : Easy to learn how to use | 250 | 265
  Autoinjector : Easy to hold in hand: number analyzed (Number of participant visits) | 253 | 281
  Autoinjector : Easy to hold in hand | 247 | 267
  Autoinjector : Easy to inject my dose: number analyzed (Number of participant visits) | 253 | 281
  Autoinjector : Easy to inject my dose | 245 | 265
  Autoinjector : Easy to know dose is complete: number analyzed (Number of participant visits) | 253 | 281
  Autoinjector : Easy to know dose is complete | 241 | 261
  Autoinjector : Easy store device in fridge: number analyzed (Number of participant visits) | 247 | 278
  Autoinjector : Easy store device in fridge | 230 | 256
  Autoinjector : Easy to remove needle shield: number analyzed (Number of participant visits) | 253 | 281
  Autoinjector : Easy to remove needle shield | 250 | 268
  Autoinjector : Easy to pickup: number analyzed (Number of participant visits) | 253 | 281
  Autoinjector : Easy to pickup | 251 | 271
  Autoinjector : Overall, easy to use: number analyzed (Number of participant visits) | 253 | 281
  Autoinjector : Overall, easy to use | 251 | 262
  Autoinjector : Dvc is stable against skin: number analyzed (Number of participant visits) | 253 | 281
  Autoinjector : Dvc is stable against skin | 244 | 264
  Autoinjector : Confident in ability to use: number analyzed (Number of participant visits) | 253 | 281
  Autoinjector : Confident in ability to use | 247 | 260
  Autoinjector : Confident my dose is complete: number analyzed (Number of participant visits) | 253 | 281
  Autoinjector : Confident my dose is complete | 244 | 263

ADVERSE EVENTS:
Time Frame: Up to 421 days
Description: All randomized participants. There were 6 participants in the 120 mg open label arm who discontinued after receiving loading dose of 240mg, these participants were moved to 240mg arm for AE analysis.
  Per protocol, AE analysis was planned per treatment regimen received.
Groups:
- Galcanezumab 120 mg - Open Label Phase: Participants received a loading dose of 240 mg galcanezumab at first dosing visit followed by 120 mg Galcanezumab once a month by subcutaneous injection for 11 months.
- Galcanezumab 240 mg - Open Label Phase: Participants received 240 mg of galcanezumab once a month by subcutaneous injection for 12 months.
- Galcanezumab 120 mg - Post-treatment Phase; Galcanezumab 240 mg - Post-treatment Phase: Participants did not receive any intervention.
Arm/Group | Galcanezumab 120 mg - Open Label Phase | Galcanezumab 240 mg - Open Label Phase | Galcanezumab 120 mg - Post-treatment Phase | Galcanezumab 240 mg - Post-treatment Phase
All-Cause Mortality (participants affected / at risk) | 0/129 | 0/141 | 0/112 | 0/124
Serious Adverse Events (participants affected / at risk) | 3/129 | 7/141 | 3/112 | 2/124
Other Adverse Events (participants affected / at risk) | 76/129 | 83/141 | 6/112 | 8/124
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Galcanezumab 120 mg - Open Label Phase (N=129) | Galcanezumab 240 mg - Open Label Phase (N=141) | Galcanezumab 120 mg - Post-treatment Phase (N=112) | Galcanezumab 240 mg - Post-treatment Phase (N=124)
Diverticulum intestinal (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Endocarditis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infective aneurysm (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Subarachnoid haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lumbar radiculopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pineal gland cyst (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemorrhagic ovarian cyst (Reproductive system and breast disorders) | 0/104 (0) | 0/119 (0) | 1/91 (1) | 0/106 (0) — All randomized female participants. There were 6 female participants in the 120 mg arm who discontinued after receiving loading dose of 240mg, these participants were moved to 240mg arm for AE analysis
Uterine leiomyoma embolisation (Surgical and medical procedures) | 0/104 (0) | 1/119 (1) | 0/91 (0) | 0/106 (0) — All randomized female participants. There were 6 female participants in the 120 mg arm who discontinued after receiving loading dose of 240mg, these participants were moved to 240mg arm for AE analysis
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Galcanezumab 120 mg - Open Label Phase (N=129) | Galcanezumab 240 mg - Open Label Phase (N=141) | Galcanezumab 120 mg - Post-treatment Phase (N=112) | Galcanezumab 240 mg - Post-treatment Phase (N=124)
Nausea (Gastrointestinal disorders) | 10 (11) | 9 (15) | 1 (1) | 0 (0)
Injection site bruising (General disorders) | 5 (5) | 8 (10) | 0 (0) | 0 (0)
Injection site erythema (General disorders) | 9 (20) | 9 (19) | 0 (0) | 0 (0)
Injection site pain (General disorders) | 22 (148) | 28 (272) | 0 (0) | 0 (0)
Injection site reaction (General disorders) | 15 (48) | 13 (32) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 8 (9) | 8 (8) | 1 (1) | 1 (1)
Sinusitis (Infections and infestations) | 14 (16) | 13 (17) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 9 (10) | 21 (23) | 0 (0) | 1 (2)
Viral upper respiratory tract infection (Infections and infestations) | 21 (27) | 16 (19) | 0 (0) | 2 (2)
Weight increased (Investigations) | 7 (7) | 4 (4) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 (12) | 8 (10) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 12 (15) | 15 (18) | 2 (2) | 3 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 8 (9) | 3 (4) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 5 (7) | 9 (11) | 0 (0) | 0 (0)
Prostatitis (Reproductive system and breast disorders) | 0/25 (0) | 0/22 (0) | 0/21 (0) | 1/18 (1) — All randomized male participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2015-09-23): https://cdn.clinicaltrials.gov/large-docs/87/NCT02614287/Prot_000.pdf
  • Statistical Analysis Plan (2015-11-23): https://cdn.clinicaltrials.gov/large-docs/87/NCT02614287/SAP_001.pdf